CLINICAL TRIAL: NCT05900180
Title: Pediatric Speech Therapy Session Frequency and Speech Outcomes
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Connecticut Children's Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22-160
Record Dates: First submitted 2023-04-20; First posted 2023-06-12 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-05

CONDITIONS: Speech Therapy; Language Disorders in Children; Articulation Disorders in Children; Communication Disorder, Childhood; Pediatric; Mode of Therapy; Frequency of Therapy
MeSH Terms: conditions — Communication Disorders | interventions — Speech Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Every-other-week therapy with home programming (Active Comparator): Receipt of standard speech therapy care (every-other-week) for 8.0 sessions
  Interventions: Behavioral: Speech Therapy
- Weekly therapy with home programming (Experimental): Receipt of speech therapy care (every week) for 8.0 sessions
  Interventions: Behavioral: Speech Therapy

INTERVENTIONS:
Behavioral: Speech Therapy — Delivery of speech therapy services

SUMMARY:
The goal of this clinical trial is to compare speech therapy outcomes in children ages 18 months to 16 years who participate in weekly speech therapy with home programming versus every-other week speech therapy with home programming in outpatient speech therapy. The main question it aims to answer is: Does a change in how often speech therapy sessions are delivered show an increased benefit in language and articulation standardized test scores? Participants will be randomly assigned to either (1) weekly or (2) every-other-week speech therapy for a total of 8 sessions. Researchers will compare these two groups to see if there are differences in speech outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Medical order for speech therapy
* Patients eligible for speech therapy at Connecticut Children's (qualify for receptive, expressive language and/or articulation therapy)
* Diagnosis of communication disorder.ICD-10 codes will be utilized pertaining to expressive, receptive language and articulation disorders (ICD-10 code specific to patient: F80.0, F80.1, F80.2, F80.4, F80.9, R47.89, R41.841)
* Patient recommended for individual (i.e. not group) treatment
* 18 months to 16 years of age
* Completed 1 plan of care (POC) with a duration of 8 sessions
* Attended at least 80% of scheduled visits during their plan of care period (still completing 8 sessions of therapy, may have extended time to completion).
* Services for a full 8-session plan of care.

Exclusion Criteria:

* - Seeking speech therapy care for treatment of disorders related to diagnosis of voice, feeding, fluency, and/or cognition
* Patient unable to complete standardized tests (EOWPVT-4, ROWPVT-4, GFTA-3, REEL-4)
* Patients in group speech therapy
* Patients younger than 18 months or older than 16 years of age
* Not willing to complete a full POC (8 sessions)
* Unable/unwilling to attend 80% of scheduled visits

Ages: 18 Months to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 39 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2027-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in Articulation and intelligibility | Baseline, immediately after treatment (up to 4 months)
  Scores on the following standardized measures: Goldman Fristoe Test of Articulation- Third Edition (GFTA-3) ; Average Standard Score range is from 86-114; an increase in standard score indicates improvement in intelligibility.
Change in Receptive vocabulary skills | Baseline, immediately after treatment (up to 4 months)
  Scores on the following standardized measure: Receptive One Word Picture Vocabulary Test- Fourth Edition (ROVPVT-4); Average Standard Score range is from 85-115; an increase in standard score indicates improvement in understanding vocabulary.
Change in Expressive vocabulary skills | Baseline, immediately after treatment (up to 4 months)
  Scores on the following standardized measure: Expressive One Word Picture Vocabulary Test- Fourth Edition (EOWPVT-4); Average Standard Score range is from 85-115; an increase in standard score indicates improvement in understanding or labeling vocabulary.
Change in Receptive and expressive early language skills | Baseline, immediately after treatment (up to 4 months)
  Scores on the following standardized measures: Receptive-Expressive Emergent Language Scale- Fourth Edition (REEL-4); Average Standard Score range is from 90-109; an increase in standard score indicates improvement in language ability score.

SECONDARY OUTCOMES:
Home Exercise Plan (HEP) provision | up to 4 months
  Parent-reported compliance with home therapy programming

CONTACTS AND LOCATIONS:
Overall Officials: Virginia Van Epps, M.Ed., Principal Investigator — Connecticut Children's Medical Center; Mary Dortenzio, MS, Study Director — Connecticut Children's Medical Center; Jodi Urzua, MS, Study Director — Connecticut Children's Medical Center; Emma Mendillo, MA, Study Director — Connecticut Children's Medical Center; Morgan Daur-Schierholz, MS, Study Director — Connecticut Children's Medical Center
Locations (1):
- Connecticut Children's Medical Center, Hartford, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No